CLINICAL TRIAL: NCT01832896
Title: A Multicenter, Open-Label Study to Assess the Tolerability and Safety of a Single, Subcutaneous Administration of Ecallantide in Children and Adolescents With Hereditary Angioedema
Brief Title: Study to Assess the Tolerability and Safety of Ecallantide in Children and Adolescents With Hereditary Angioedema
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI indicated departure from institution, inability to complete study.
Sponsor: NYU Langone Health (Other)
Collaborators: Dyax Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DX-88/IST-5
Record Dates: First submitted 2013-04-04; First posted 2013-04-16 (Estimated); Last update posted 2023-03-31 (Actual); Status verified 2017-01

CONDITIONS: Hereditary Angioedema Types I and II
Keywords: Hereditary Angioedema; Children; Adolescents; Ecallantide
MeSH Terms: conditions — Hereditary Angioedema Types I and II; Angioedemas, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ecallantide (Experimental): Study Medication, Dose, and Mode of Administration:
  Single dose of ecallantide subcutaneous dosing:
  * Age less than 10: Weight <25 Kg: 10mg subcutaneously at one site; 25-50kg: 20mg subcutaneously, 10mg per site for 2 separate sites; >50 kg 30mg subcutaneously, 10mg per site for 3 separate sites. Dosing will not exceed 30mg.
  * Age greater than 10: 10mg per site for 3 separate sites. Dosing will not exceed 30mg.
  Interventions: Drug: Ecallantide subcutaneous dosing

INTERVENTIONS:
Drug: Ecallantide subcutaneous dosing — For acute attacks of Hereditary Angioedema in children and adolescents, Ecallantide will be administered.

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of a single Subcutaneous (SC) dose of Ecallantide in children and adolescents with Hereditary Angioedema (HAE).

DETAILED DESCRIPTION:
This pilot study is an open-label, non-randomized, single-arm study to evaluate the tolerability and safety of a single SC administration of ecallantide in up to approximately 10 pediatric subjects with HAE during an initial acute attack. The study is planned to enroll subjects 2 through 15 years of age who present with an acute cutaneous, abdominal, or laryngeal HAE attack. No more than 3 study sites will be included until a goal of 10 patients is achieved.

After treatment for an initial attack, one additional open label treatment with ecallantide will be offered to subjects contingent upon having been treated previously and presenting with a subsequent acute cutaneous, abdominal, or laryngeal attack of HAE at least 7 days after initial treatment. Open-label treatment for a second HAE attack will continue until 10 patients have been treated for an initial attack. Safety evaluations will be performed at each subsequent ecallantide-treated attack as for the initial treated attack

ELIGIBILITY:
Inclusion Criteria:

1. 2 through 15 years of age, inclusive (ie, from the second birthday through the day prior to the sixteenth birthday) at the time of the subject's first attack.
2. Documented diagnosis of HAE type I or II. Diagnosis must be confirmed by a documented immunogenic (below the lower limit of normal) and/or functional (< 50% of normal levels) C1- Inhibitor deficiency. Diagnosis may be on the basis of historic data or by diagnostic testing conducted at the time of screening.
3. Informed consent (and subject assent as appropriate) signed by the subject's parent(s) or legal guardian(s).

Exclusion Criteria:

1. History of an adverse reaction (AE) to Ecallantide in the past
2. Diagnosis of angioedema other than HAE
3. Participation in another clinical study during the 30 days prior to treatment
4. Any known factor/disease that might interfere with the treatment compliance, study conduct, or result interpretation
5. Congenital or acquired cardiac anomalies that interfere significantly with cardiac function.
6. Treatment with angiotensin converting enzyme (ACE) inhibitors within 7 days prior to treatment.
7. Use of hormonal contraception within the 90 days prior to treatment for females of childbearing potential
8. The subject is pregnant or breastfeeding

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Measurement of time to symptomatic improvement from acute attacks of hereditary angioedema | 28 days
  Time to symptom relief. Time to minimal symptoms. An improvement assessment will also be performed at each of the following timepoints: pre -treatment, every 30 minutes for the first 2 hours and then hourly through discharge and at the 28 day clinic visit.
  Incidence of need for rescue medication. Incidence of worsening despite use of ecallantide.

SECONDARY OUTCOMES:
Number of Partcipants with Adverse Events | 28 Days
  Study Partcipants will be monitored for adverse events, changes in laboratory values, physical exam, vital sign changes and ECG changes. Vital signs, including body temperature, heart rate and sitting blood pressure, will be assessed at screening, Pre-treatment, every 30 minutes for the first 2 hours and then hourly through discharge and at the 28 day clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Davis-Lorton, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop-University Hosptial Clinical Trials Center, Mineola, New York, United States